CLINICAL TRIAL: NCT06059573
Title: The Accuracy of Dental Implant Placement Using Robotic System-assisted Surgery and Freehand Surgery: a Randomized Clinical Trial
Brief Title: The Accuracy of Dental Implant Placement Using Robotic System-assisted Surgery and Freehand Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qi Yan (Other)
Responsible Party: Sponsor-Investigator, Qi Yan, associate professor, Hospital of Stomatology, Wuhan University
Organization: Hospital of Stomatology, Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022[07]
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dental Implant
Keywords: robot-guided surgery; freehand; dental implant robot; accuracy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-guided (Experimental): Implant placement by robot-guided based on a digital plan
  Interventions: Procedure: dental implant robot
- Freehand surgery (Active Comparator): Implant placement by freehand based on a digital plan
  Interventions: Procedure: Freehand surgery

INTERVENTIONS:
Procedure: dental implant robot — Implant placement will be navigated by a dental implant robot based on a digital plan.
  Arms: Robot-guided
Procedure: Freehand surgery — Implant will be placed under freehand surgery.
  Arms: Freehand surgery

SUMMARY:
We plan to conduct this randomized clinical trial to compare the implant positional accuracy of robotic system-assisted implant surgery with that of conventional freehand implant surgery. Patients will be enrolled and randomly assigned to either an experimental group that underwent robotic surgery or a control group that underwent freehand surgery, to evaluate the accuracy of implant in both groups.

DETAILED DESCRIPTION:
Oral implants have become a widely used treatment modality for patients with missing or edentulous teeth. Previous studies have shown that implant accuracy is associated with implant success and long-term outcomes. Therefore, we plant to conduct this randomized clinical trial to compare the implant positional accuracy of robotic system-assisted implant surgery with that of conventional freehand implant surgery. Patients will be enrolled and randomly assigned to either an experimental group that underwent robotic surgery or a control group that underwent freehand surgery. By comparing the preoperative planned implant position with the actual postoperative implant position using CBCT, we will evaluate the accuracy of implant in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Single missing teeth with adjacent and opposing healthy natural teeth;
2. Healthy patients;
3. Sufficient alveolar bone available for implant placement.

Exclusion Criteria:

1. Pregnancy or intention to become pregnant at any point during the study duration
2. With any systemic diseases/conditions that are contraindications to dental implant...

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-10-07 (Estimated); Primary Completion 2023-11-07 (Estimated); Study Completion 2023-12-07 (Estimated)

PRIMARY OUTCOMES:
Implant positional accuracy | immediately after surgery
  Implant accuracy will be measured as distance discrepancy at implant platform and implant apex, and angular discrepancy of implant axis between the digital plan and the actual position of the implant assessed digitally at the end of the procedure. Pre- and post-operative CBCT will be used for measurement.

SECONDARY OUTCOMES:
Surgery complication | Immediately and seven days after surgery
  Complication related to implant placement surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Yan, PhD, Principal Investigator — School & Hospital of Stomatology, Wuhan University; Yufeng Zhang, PhD, Study Chair — School & Hospital of Stomatology, Wuhan University
Locations (1):
- School & Hospital of Stomatology, Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No